CLINICAL TRIAL: NCT02482207
Title: A Randomized, Double-blind, Active-controlled Study to Assess the Effect of Rosuvastatin on Coronary Flow Reserve in Hypertensive Patients With Cardiovascular Risk
Brief Title: Effect of Rosuvastatin on Coronary Flow Reserve in Hypertensive Patients With Cardiovascular Risk
Acronym: RESERVE II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-0610
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 10 mg qd for 1 year and life style modification
  Interventions: Drug: Rosuvastatin; Behavioral: Life style modification
- Placebo (Placebo Comparator): Life style modification alone
  Interventions: Behavioral: Life style modification

INTERVENTIONS:
Drug: Rosuvastatin
  Arms: Rosuvastatin
Behavioral: Life style modification

SUMMARY:
Investigators recently demonstrated that coronary flow reserve (CFR) significantly improved after rosuvastatin therapy in hypertensive patients with average levels of serum cholesterol by measuring the change in CFR after 1 year treatment with rosuvastatin in the RESERVE (Rosuvastatin Effect on Coronary Flow Reserve in Hypertensive Patients) I trial. However, the absence of a placebo group made it difficult to exclude the possibility that lifestyle modification and antihypertensive medication also played a role in improving CFR in our previous study. In a double-blind, randomized trial, investigators try to examine the hypothesis that rosuvastatin added to lifestyle modification will be superior to lifestyle modification alone in improving CFR in hypertensive patients .

DETAILED DESCRIPTION:
Statin therapy improves coronary flow reserve (CFR) and decreases cardiac morbidity and mortality in patients with coronary artery disease (CAD) and hypercholesterolemia via pleiotropic effects of statins, including regression of atheroma, stabilization of atherosclerotic plaques. Lipid lowering with a statin also provided beneficial effects in hypertensive patients with average levels of serum total cholesterol in the Anglo-Scandinavian Cardiac Outcomes Trial-Lipid Lowering Arm (ASCOT-LLA). Improvements in endothelial dysfunction and CFR may be related to the beneficial effects of statins in hypertensive patients without hypercholesterolemia.

Previously CFR could be invasively measured using a Doppler guide wire in a cardiac catheterization laboratory, but recent advances in echocardiographic imaging techniques have made it feasible to measure CFR noninvasively in patients without CAD, which highly correlates with the CFR measured by invasive means.Accordingly, investigators recently demonstrated that CFR significantly improved after rosuvastatin therapy in hypertensive patients with average levels of serum cholesterol by measuring the change in CFR after 1 year treatment with rosuvastatin and also found a weak correlation between the change of CFR and the change of LDL cholesterol in the RESERVE (Rosuvastatin Effect on Coronary Flow Reserve in Hypertensive Patients) I trial. However, this trial could not include placebo-control group due to the limited study budget. Although CFR was measured by blinded, batch reading of stored echocardiographic images, bias in measurement might affect the result. In our previous study, study patients continued taking their antihypertensive medications and were educated to follow lifestyle modification during the study period, which may have influenced the change in CFR during follow-up, and the absence of a placebo group made it difficult to exclude the possibility that lifestyle modification and antihypertensive medication also played a role in improving CFR. Investigators hypothesize that rosuvastatin added to lifestyle modification will be superior to lifestyle modification alone in improving CFR in controlled hypertensive patients with cardiovascular risk, and try to examine this hypothesis in a double-blind, randomized comparison study using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Controlled Hypertension: treated SBP<140 mmHg and DBP<90 mmHg with angiotensin receptor blocker (ACE inhibitor) and/or calcium channel blocker LDL cholesterol ≥ 130mg/dL
* Patients with statin-naive state, defined as receiving no statin therapy for more than 6 months during the previous 12 months.
* Any 1 of these cardiovascular risk factors required: smoking, age over 55 (men) or 65 (women), history of cerebrovascular event, family history of early coronary heart disease before age 55, HDL cholesterol < 40 mg/dL
* The patient agrees to the study protocol and the schedule of clinical and echocardiographic follow-up, and provides informed, written consent, as approved by the Institutional Review Board

Exclusion Criteria:

* A previous history of intolerance or hypersensitivity to statins
* Uncontrolled hypertension; SBP≥140 mmHg or DBP≥90 mmHg
* Previous myocardial infarction or currently treated angina pectoris
* Stroke, transient ischemic attack < 3 months
* Secondary hypertension
* Diabetes mellitus
* Peripheral vascular disease
* Fasting serum triglyceride > 500 mg/dL
* Clinical congestive heart failure
* Uncontrolled arrhythmia
* Left ventricular hypertrophy: LV mass index >134g/m2 (male) or >110g/m2 (female)
* Concomitant clinically important hematological, gastrointestinal, hepatic, renal or other disease
* Pregnant or lactating women and those of child-bearing potential
* Unwillingness or inability to comply with the procedures described in this protocol

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Difference of Coronary flow velocity reserve | 1 year follow-up
  Averaged value of coronary flow velocity reserve will be obtained at 1 year follow-up

SECONDARY OUTCOMES:
Change of coronary flow velocity reserve | 1 year follow-up
  Change of coronary flow velocity reserve from baseline to 1 year follow-up
Change of LDL cholesterol | 1 year follow-up
  Change of LDL cholesterol from baseline to 1 year follow-up
Change of C reactive protein (CRP) | 1 year follow-up
  Change of CRP from baseline to 1 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun BJ, Hwang E, Jang JY, Kim DH, Song JM, Kang DH. Effect of rosuvastatin on coronary flow reserve in patients with systemic hypertension. Am J Cardiol. 2014 Oct 15;114(8):1234-7. doi: 10.1016/j.amjcard.2014.07.046. Epub 2014 Jul 30. PMID 25159238